CLINICAL TRIAL: NCT00798824
Title: The Impact of Nasogastric Indwelling Versus Oral Intermittent Tube Feeding Methods on Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Judy Kublick, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B2008:072
Record Dates: First submitted 2008-09-12; First posted 2008-11-26 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Premature Infants
Keywords: tube feeding; premature infant
MeSH Terms: conditions — Premature Birth | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indwelling nasogastric tube placement (Active Comparator)
  Interventions: Procedure: Indwelling nasogastric tube placement; Device: Nasogastric tube
- Intermittent orogastric tube placement (Active Comparator)
  Interventions: Procedure: Intermittent orogastric tube placement; Device: Oral gastric tube

INTERVENTIONS:
Procedure: Indwelling nasogastric tube placement — The premature infant is fed with an indwelling nasogastric tube during feeding transition.
  Other Names: Nasogastric tube
  Arms: Indwelling nasogastric tube placement
Procedure: Intermittent orogastric tube placement — The premature infant is fed with an intermittently placed orogastric tube during feeding transition.
  Other Names: Oral gastric tube
  Arms: Intermittent orogastric tube placement
Device: Nasogastric tube — Premature infants will be fed with a nasogastric tube in place and their feeding behaviors will be noted till discharge.
  Arms: Indwelling nasogastric tube placement
Device: Oral gastric tube — Premature infants will be fed with intermittent orogastric tube placement and their feeding behaviors will be noted till discharge.
  Arms: Intermittent orogastric tube placement

SUMMARY:
This clinical pilot trial is being conducted to learn more about the infant's feeding behavior while being fed by indwelling nasogastric tube placement or by intermittent oral tube placement.

Healthy preterm infants who are transitioning from gavage to oral feedings via oral intermittent tube insertion may achieve full oral feeds by bottle/breast at an earlier gestational age than infants feeding with indwelling tubes and may be ready for earlier discharge.

DETAILED DESCRIPTION:
Independent feeding is often one of the last competencies that the premature infant must accomplish prior to discharge from hospital. Feeding is a complex task for the premature infant to accomplish and it often takes many weeks for the infant to learn how to feed. Therefore, tube feeding is required for the infant to ingest adequate nutrition during the transition from gavage feeding to oral feeding. Both intermittent oral gavage tube placement and indwelling nasogastric tube placement are acceptable methods for feeding preterm infants. However, it is not known which tube feeding method will support an expedited transition to oral feeding. The choice of using one method over the other is currently based on the individual health care provider's opinion or historical institutional practices and insufficient evidence is available to guide tube feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born between 30-33 and 6/7th weeks gestation are an appropriate size for gestational age, are not on Oxygen are of any race, sex and require tube feeding and are less than 34 and 3/7th weeks gestation.

Exclusion Criteria:

* infants with neurological abnormalities or insults, IVH greater than a grade of two, PVL, birth asphyxia, seizures, cord has less than 7.0 ph, chest compressions, infants who require abstinence scoring, infants with major congenital anomalies or major genetic anomalies that impact feeding ability such as diaphragmatic hernia and cleft palate, major cardiac defects, infants who develop necrotizing enterocolitis, infants who received more than 14 days of intubation or CPAP or oxygen by nasal prongs and infants of diabetic or alcoholic mothers.

Ages: 30 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Gestational age of the last required tube feed. | Last required tube feed

SECONDARY OUTCOMES:
Discharge date | Discharge date
The amount suckled per day | Discharge date

CONTACTS AND LOCATIONS:
Overall Officials: Judy A Kublick, Grad student, Principal Investigator — University of Manitoba
Locations (1):
- Intermediate Care Unit, Health Sciences Centre, Winnipeg, Manitoba, Canada